CLINICAL TRIAL: NCT07304440
Title: Adia MED of Winter Park LLC Autism Spectrum Disorder Research Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adia Med of Winter Park LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Adia Med ASD Research Study
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Autism Spectrum Disorder; Autism; ASD; Autism Spectrum Disorder (ASD)
Keywords: Glutathione; Intravenous glutathione; Glutathione therapy; Antioxidant therapy; Oxidative stress; Immune modulation; Anti-inflammatory therapy; Autism; Autism Spectrum Disorder; ASD; Autism symptoms; Stem cell therapy; MSCs; Mesenchymal stem cells; Regenerative medicine; Cellular therapy; Hematopoietic stem cells (HSCs); Allogeneic stem cells
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Glutathione

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glutathione with Stem Cells (Experimental)
  Interventions: Biological: Umbilical Cord Blood-Derived Stem Cells and Exosomes; Drug: Glutathione
- Glutathione Only (Active Comparator)
  Interventions: Drug: Glutathione

INTERVENTIONS:
Biological: Umbilical Cord Blood-Derived Stem Cells and Exosomes — Intravenous infusion of cryopreserved allogeneic umbilical cord blood-derived product containing viable mononuclear cells (including hematopoietic and mesenchymal stem/stromal cells) and exosomes.
  Arms: Glutathione with Stem Cells
Drug: Glutathione — Reduced L-glutathione administered Intravenous infusion once monthly for 3 months (Phase I)

SUMMARY:
This 24-month study is testing whether adding AdiaVita, an umbilical cord blood-derived stem cell and exosome product, to glutathione therapy helps improve autism symptoms in children ages 3-12 more than glutathione alone. Children will be randomly placed into one of two groups for the first three months: one group receives glutathione only, and the other receives glutathione plus monthly intravenous AdiaVita infusions. Both groups also use topical glutathione cream twice daily at home. Autism symptoms will be tracked over two years using the Autism Treatment Evaluation Checklist (ATEC) filled out by parents and by therapists or teachers. Safety, side effects, quality of life, and overall well-being will be closely monitored through regular clinic visits, physical exams, blood tests, and adverse event reporting. After the initial three-month phase, children who received glutathione alone may cross over to receive AdiaVita infusions at no additional cost if safety checks at month 6 are satisfactory. Approximately 100 children with a confirmed autism diagnosis from the Central Florida area will take part. Participation is completely voluntary, and families may withdraw at any time.

DETAILED DESCRIPTION:
This study evaluates the safety and preliminary effectiveness of AdiaVita, an umbilical cord blood-derived stem cell and exosome product, when combined with glutathione for improving symptoms of Autism Spectrum Disorder in children ages 3-12. Participants are randomized to receive either glutathione alone or glutathione plus AdiaVita during the initial three-month treatment phase. Symptoms are measured using repeated Autism Treatment Evaluation Checklist assessments completed by both parents and therapists/teachers throughout the 24-month follow-up period. The primary outcome is change in total ATEC scores at Month 6, with secondary outcomes including safety, tolerability, quality of life, and overall wellness. Children in the glutathione-only group may enter a Phase II extension in which they later receive stem cell infusions at no additional cost if safety requirements are met at the six-month interim review. All clinical visits include physical exams, vitals, adverse event reviews, and post-infusion monitoring. Treatments involve monthly intravenous administration and twice-daily at-home topical glutathione during Phase One. Blood tests are completed prior to key visits to ensure medical stability, and serious adverse events trigger immediate medical attention and reporting. Risks include infusion-related discomfort, headache, fever, allergic reactions, or rare immune responses, with theoretical long-term risks noted. Potential benefits include improvement in social interaction, communication, and behavioral symptoms, although no benefits are guaranteed. Participation is voluntary and families may withdraw at any time, though study costs already paid are non-refundable. Data are stored securely with coded identifiers and only authorized parties may access identifiable information. Recruitment occurs through direct contact, clinic advertising, community outreach, and social media. Approximately 100 children Nation Wide are expected to participate and must have a confirmed ASD diagnosis prior to enrollment. Exclusion criteria include severe allergies to the study products, uncontrolled medical conditions, and recent participation in another interventional trial. No monetary incentives are offered, and families instead pay a fixed fee of $12,000 for Phase One, which covers all procedures and also includes Phase II if applicable. Outcomes will contribute to scientific knowledge regarding the safety and possible clinical utility of stem cell-based therapies for ASD.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-12 years
* Confirmed ASD diagnosis (DSM-5 criteria, supported by ADOS-2)
* Parent/guardian willingness to consider experimental treatments and comply with study requirements
* Ability to attend all scheduled visits

Exclusion Criteria:

* Severe allergies to study products
* Significant uncontrolled medical conditions
* Pregnancy or breastfeeding (if applicable)
* Participation in another interventional trial within 30 days

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Total Autism Treatment Evaluation Checklist (ATEC) Score at Month 6 | Baseline and Month 6
  The Autism Treatment Evaluation Checklist (ATEC) is a caregiver-completed questionnaire designed to evaluate treatment effectiveness in autism by assessing symptoms across four domains (Speech/Language/Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). Total ATEC scores range from 0 to 180, with higher scores indicating greater severity of autism symptoms (worse outcome) and lower scores indicating fewer symptoms (better outcome).

SECONDARY OUTCOMES:
Change from Baseline in Total Autism Treatment Evaluation Checklist (ATEC) Score at Month 3 | Baseline and Month 3
  The Autism Treatment Evaluation Checklist (ATEC) is a caregiver-completed questionnaire designed to evaluate treatment effectiveness in autism by assessing symptoms across four domains (Speech/Language/Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). Total ATEC scores range from 0 to 180, with higher scores indicating greater severity of autism symptoms (worse outcome) and lower scores indicating fewer symptoms (better outcome).
Change from Baseline in Total Autism Treatment Evaluation Checklist (ATEC) Score at Months 12 and 24 | Baseline, Month 12, and Month 24
  The Autism Treatment Evaluation Checklist (ATEC) is a caregiver-completed questionnaire designed to evaluate treatment effectiveness in autism by assessing symptoms across four domains (Speech/Language/Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). Total ATEC scores range from 0 to 180, with higher scores indicating greater severity of autism symptoms (worse outcome) and lower scores indicating fewer symptoms (better outcome).
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events | Baseline through Month 24

CONTACTS AND LOCATIONS:
Locations (1):
- Adia Med Of Winter Park, Winter Park, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided